CLINICAL TRIAL: NCT07294664
Title: Clinical Study of SHR1701 in Combination With CAPOX and SHR2554 for First-line Treatment of Advanced Gastric Cancer
Brief Title: PD1/TGFβ In Combination With EZH2 And Chemotherapy For First - Line Treatment Of Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yongxu Jia, Chief Investigator, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-022
Record Dates: First submitted 2025-07-30; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Gastric Cancer; SHR1701
MeSH Terms: interventions — SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1701+SHR2554+CAPOX (Experimental)
  Interventions: Drug: SHR1701; Drug: SHR2554; Drug: CAPOX

INTERVENTIONS:
Drug: SHR1701 — SHR1701:1800mg,d1,Q3W
Drug: SHR2554 — SHR2554 350mg,bid
Drug: CAPOX — Capecitabine:1000mg/kg,bid,d1-d14,Q3W Oxaliplatin:130mg/2,d1,Q3W

SUMMARY:
Immunotherapy combined with chemotherapy has become the standard first-line treatment regimen for gastric cancer. However, a subset of patients still fail to benefit or derive only limited benefit from this approach. This study aims to evaluate the addition of an EZH2 inhibitor with immunomodulatory functions to the foundation of immunotherapy plus chemotherapy, with the goal of further enhancing treatment benefit for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily agree to participate in this study and sign the informed consent form;
2. Age ≥ 18 years;
3. ECOG PS score 0-1;
4. Pathologically confirmed adenocarcinoma of the stomach/gastroesophageal junction;
5. Clinical staging based on contrast - enhanced CT/MRI (with endoscopic ultrasound and diagnostic laparoscopy if necessary). Patients with stage III-IV (8th edition of the AJCC Gastric Cancer TNM Staging) non - resectable locally advanced or metastatic disease; the feasibility of curative surgery for patients is determined by multidisciplinary team (MDT) discussion;
6. Patients who have not previously received systemic therapy for advanced disease;Note: Neoadjuvant therapy is not counted as a line of therapy. If recurrence occurs within 6 months after completion of adjuvant therapy, the adjuvant therapy is defined as first - line therapy. If recurrence occurs more than 6 months after completion of adjuvant therapy, the adjuvant therapy is not counted as a line of therapy.
7. Have measurable lesions meeting Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
8. Subjects' baseline blood routine and biochemical indices meet the following criteria (no blood transfusion/blood products received, and no granulocyte colony - stimulating factor (G - CSF) or other hematopoietic growth factors used for correction within 14 days before the first dose):

   Hemoglobin ≥ 90 g/L; Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelets ≥ 80×10^9/L; ALT, AST ≤ 2.5 × upper limit of normal (ULN); if the patient has liver metastasis, ALT and AST ≤ 5 × ULN; Serum total bilirubin ≤ 1.5 × ULN; Serum creatinine (Cr) ≤ 1.5 × ULN or estimated creatinine clearance > 50 mL/min (For males: Creatinine clearance = ((140 - age) × weight) / (72 × serum Cr); For females: Creatinine clearance = ((140 - age) × weight) / (72 × serum Cr) × 0.85; Weight unit: kg; Serum Cr unit: mg/mL); Serum albumin ≥ 30 g/L;
9. No serious concurrent diseases that would result in a life expectancy of < 5 years
10. Female subjects of childbearing potential must undergo a serum pregnancy test within 72 hours prior to the first dose, with a negative result, and agree to use highly effective methods of contraception during treatment and for 90 days after the end of treatment. For male subjects whose partners are female of childbearing potential, they must agree to use highly effective methods of contraception during treatment and for 90 days after the end of treatment.
11. Agree to provide blood and/or histological specimens.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Known HER2 positivity;
3. Patients with adverse events from previous treatments (except alopecia) that have not resolved to ≤ Grade 1 (CTCAE v5.0);
4. History of other malignant diseases within the past 5 years or concurrent malignant diseases, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
5. History of uncontrolled epilepsy, central nervous system diseases, or mental disorders, where the investigator judges that the clinical severity may hinder the signing of informed consent or affect the patient's adherence to oral medications;
6. Clinically significant (i.e., active) heart disease that is not well-controlled, such as: (1) Symptomatic coronary heart disease; (2) New York Heart Association (NYHA) Class II or worse congestive heart failure or severe arrhythmias requiring medication intervention; (3) Myocardial infarction within the past 12 months; (4) QTc interval ≥ 450 ms in males or ≥ 470 ms in females; (5) Left ventricular ejection fraction (LVEF) < 50%;
7. Arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, pulmonary embolism, etc.;
8. Clinically significant bleeding symptoms or definite bleeding tendency within 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc. If fecal occult blood is positive during screening, a re-examination is allowed; if still positive after re-examination, gastroscopy may be performed as clinically indicated (except those who have undergone gastroscopy within 3 months before enrollment to rule out such conditions);
9. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., patients with hemophilia, coagulopathy, thrombocytopenia, etc.);
10. Patients with upper gastrointestinal obstruction, abnormal physiological function, or malabsorption syndrome that may affect the absorption of oral medications; patients with a history of gastrointestinal perforation, intra-abdominal abscess, or intestinal obstruction within the past 3 months, or with imaging findings/clinical symptoms suggesting concurrent intestinal obstruction;
11. Abnormal coagulation function (INR > 2.0 or prothrombin time > 16 seconds), with bleeding tendency or receiving thrombolytic or anticoagulant therapy (prophylactic use of low-dose aspirin, low-molecular-weight heparin, etc., is allowed);
12. Patients with chemotherapy-induced neurotoxicity who are judged by the investigator as unsuitable for oxaliplatin use cannot be included in Intervention Arm 1; however, patients with only deep tendon reflex (DTR) loss may not be excluded;
13. Patients who have undergone organ transplantation and require immunosuppressive therapy; patients who have used immunosuppressive drugs or systemic corticosteroids for immunosuppressive purposes within 14 days prior to the first dose (e.g., > 10 mg/day prednisone or equivalent dose of other drugs);
14. With active ulcers, unhealed wounds, or fractures;
15. Patients with hypertension that cannot be well-controlled with antihypertensive medications (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
16. Known hypersensitivity to any investigational drugs or excipients; Urinalysis indicating urinary protein ≥ ++, with confirmed 24-hour urinary protein excretion > 1.0 g;
17. Patients with clinically symptomatic serous cavity effusions (including ascites, pleural effusion, pericardial effusion) requiring symptomatic management; asymptomatic serous cavity effusion patients are allowed to enroll; patients with symptomatic serous cavity effusions that are well-controlled after active management such as drainage may be enrolled at the investigator's discretion;
18. Active hepatitis (for hepatitis B: HBsAg positive with HBV DNA ≥ 500 IU/ml; for hepatitis C: HCV antibody positive with HCV viral load > upper limit of normal); patients in active infection phase requiring antimicrobial therapy (e.g., antibacterial or antifungal treatment);
19. Currently having interstitial pneumonia or interstitial lung disease, or other conditions that may interfere with the judgment and management of immune-related pulmonary toxicity, such as pulmonary fibrosis, organizing pneumonia, pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or those with active pneumonia or severe pulmonary function impairment shown by screening CT; patients with active pulmonary tuberculosis;
20. Patients with active autoimmune diseases or a history of autoimmune diseases with potential for recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects whose condition is controllable with hormone replacement therapy may be included]); patients with skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia), type 1 diabetes mellitus controllable with insulin therapy, or those with a history of childhood asthma that has completely resolved without any intervention may be enrolled; asthmatic patients requiring bronchodilators for intervention cannot be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
ORR | assessed up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided